CLINICAL TRIAL: NCT02260700
Title: A Randomized, Open-Label, 3-Way Crossover Study in Healthy Older Male Subjects to Evaluate the Bioavailability, Food Effect, Safety and Tolerability of A Solid Dosage Formulation of JNJ-54861911
Brief Title: A Study to Evaluate Bioavailability, Food Effect, Safety and Tolerability of a Solid Dosage Formulation of JNJ-54861911 in Healthy Older Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR102380; 54861911ALZ1003 (Other: Janssen Research & Development, LLC); 2013-002650-70 (EudraCT Number)
Record Dates: First submitted 2014-10-06; First posted 2014-10-09 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
Keywords: Healthy; Bioavailability; Alzheimer's Disease; JNJ-54861911
MeSH Terms: conditions — Alzheimer Disease | interventions — atabecestat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Sequence 1 (ABC) (Experimental): Participants will receive Treatment A (single dose of JNJ-54861911 25 milligram (mg) oral suspension formulation under fasted conditions) in Period 1; followed by Treatment B (single oral dose of JNJ-54861911 25 mg solid formulation under fasted conditions) in Period 2; followed by Treatment C (single oral dose of JNJ-54861911 25 mg solid formulation under fed conditions) in Period 3. A washout period of at least 6 days will be maintained between each treatment period.
  Interventions: Drug: JNJ-54861911 (Treatment A); Drug: JNJ-54861911 (Treatment B); Drug: JNJ-54861911 (Treatment C)
- Sequence 2 (ACB) (Experimental): Participants will receive Treatment A (single dose of JNJ-54861911 25 milligram (mg) oral suspension formulation under fasted conditions) in Period 1; followed by Treatment C (single oral dose of JNJ-54861911 25 mg solid formulation under fed conditions) in Period 2; followed by Treatment B (single oral dose of JNJ-54861911 25 mg solid formulation under fasted conditions) in Period 3. A washout period of at least 6 days will be maintained between each treatment period.
  Interventions: Drug: JNJ-54861911 (Treatment A); Drug: JNJ-54861911 (Treatment B); Drug: JNJ-54861911 (Treatment C)
- Sequence 3 (BAC) (Experimental): Participants will receive Treatment B (single dose of JNJ-54861911 25 mg solid formulation under fasted conditions) in Period 1; followed by Treatment A (single oral dose of JNJ-54861911 25 milligram (mg) oral suspension formulation under fasted conditions) in Period 2; followed by Treatment C (single oral dose of JNJ-54861911 25 mg solid formulation under fed conditions) in Period 3. A washout period of at least 6 days will be maintained between each treatment period.
  Interventions: Drug: JNJ-54861911 (Treatment A); Drug: JNJ-54861911 (Treatment B); Drug: JNJ-54861911 (Treatment C)
- Sequence 4 (BCA) (Experimental): Participants will receive Treatment B (single dose of JNJ-54861911 25 mg solid formulation under fasted conditions) in Period 1; followed byTreatment C (single dose of JNJ-54861911 25 mg solid formulation under fed conditions) in Period 2; followed by Treatment A (single dose of JNJ-54861911 25 milligram (mg) oral suspension formulation under fasted conditions) in Period 3. A washout period of at least 6 days will be maintained between each treatment period.
  Interventions: Drug: JNJ-54861911 (Treatment A); Drug: JNJ-54861911 (Treatment B); Drug: JNJ-54861911 (Treatment C)
- Sequence 5 (CAB) (Experimental): Participants will receive Treatment C (single dose of JNJ-54861911 25 mg solid formulation under fed conditions) in Period 1; followed by Treatment A (single dose of JNJ-54861911 25 milligram (mg) oral suspension formulation under fasted conditions) in Period 2; followed by Treatment B (single dose of JNJ-54861911 25 mg solid formulation under fasted conditions) in Period 3. A washout period of at least 6 days will be maintained between each treatment period.
  Interventions: Drug: JNJ-54861911 (Treatment A); Drug: JNJ-54861911 (Treatment B); Drug: JNJ-54861911 (Treatment C)
- Sequence 6 (CBA) (Experimental): Participants will receive Treatment C (single dose of JNJ-54861911 25 mg solid formulation under fed conditions) in Period 1; followed by Treatment B (single dose of JNJ-54861911 25 mg solid formulation under fasted conditions) in Period 2; followed by Treatment A (single dose of JNJ-54861911 25 milligram (mg) oral suspension formulation under fasted conditions) in Period 3. A washout period of at least 6 days will be maintained between each treatment period.
  Interventions: Drug: JNJ-54861911 (Treatment A); Drug: JNJ-54861911 (Treatment B); Drug: JNJ-54861911 (Treatment C)

INTERVENTIONS:
Drug: JNJ-54861911 (Treatment A) — Participants will receive a single oral 25 mg dose of JNJ-54861911 as Treatment A (oral suspension formulation) under fasted conditions in one of the treatment periods.
Drug: JNJ-54861911 (Treatment B) — Participants will receive a single oral 25 mg dose of JNJ-54861911 as Treatment B (solid formulation) under fasted conditions in one of the treatment periods.
Drug: JNJ-54861911 (Treatment C) — Participants will receive a single oral 25 mg dose of JNJ-54861911 as Treatment C (solid formulation) under fed conditions in one of the treatment periods.

SUMMARY:
The purpose of this study is to determine pharmacokinetics (the study of the way a drug enters and leaves the blood and tissues over time) and the relative-bioavailability (the extent to which a drug or other substance becomes available to the body) of JNJ-54861911 solid dosage formulation compared with JNJ 54861911 oral suspension formulation in healthy older male participants.

DETAILED DESCRIPTION:
This is a randomized (study medication assigned to participants by chance), open-label (all people know the identity of the intervention), single-center, single-dose and 3-way Crossover (the same medications provided to all participants but in different sequence) study to determine the bioavailability of JNJ-54861911 solid dosage formulation in healthy older male participants. The study will consist of 3 parts: Screening Phase (that is, 28 days before study commences on Day 1), an open-label treatment Phase (consists of 3 single-dose treatment periods, either a single oral suspension formulation [Treatment A] or solid formulation 25 milligram (mg) dose of JNJ-54861911 under fasted [Treatment B] or fed conditions [Treatment C] in subsequent 3-treatment periods; each treatment period separated with washout period of 6 days) and follow-up Phase (7 to 14 days after last dose administration). The maximal study duration for a participant will not exceed 8 weeks. All the eligible participants will be randomly assigned to 1 of the 6 treatment sequences. Followed by an overnight fast of at least 10 hours participants will be administered with study treatment under fasted condition or fed condition (30 minutes after high-fat, high-calorie breakfast). Participants will not be allowed to have food until 4 hours of drug administration. Blood samples will be collected for evaluation of pharmacokinetics at pre-dose and post-dose of study treatment. Bioavailability will be primarily evaluated by pharmacokinetic parameters. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI; weight [kilogram(kg)]/height^2 [meter square (m^2)]) between 18 and 30 kg/m^2, (inclusive)
* Be healthy for their age group with or without medication on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at Screening or admission. Minor deviations in ECG, which are not considered to be of clinical significance to the investigator, are acceptable
* Be healthy on the basis of clinical laboratory tests performed at Screening. If the results of the serum chemistry panel [including liver enzymes], hematology, or urinalysis are outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant. This determination must be recorded in the participants' source documents and initialed by the investigator
* Men who are sexually active with a woman of childbearing potential and have not had a vasectomy must agree to use a barrier method of birth control for example, either condom with spermicidal foam/gel/film/cream/suppository or partner with occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository, and all men must also not donate sperm during the study and for 3 months after receiving the last dose of study drug. In addition, their female partners should also use an appropriate method of birth control for at least the same duration
* Participants' must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study

Exclusion Criteria:

* Participant has a clinically significant abnormal physical examination, vital signs or 12 lead ECG (including QTc greater than (>) 450msec, Left Bundle Branch Block, permanent pacemaker or implantable cardioverter defibrillator) at Screening or admission
* Participant has a history of or current liver or renal insufficiency; significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic disturbances
* Use of any prescription or over-the-counter medication, herbal medication, vitamins, or mineral supplements within 14 days prior to study drug administration (not including paracetamol). Medication for chronic use in age related disease will be allowed after approval by both the investigator and to the sponsor. No change in dose or regimen will be permitted during the study that is, from the Screening visit until the follow-up visit
* Participant has a history of spontaneous, prolonged or severe bleeding of unclear origin
* Participant has a history of epilepsy or fits or unexplained black-outs other than vasovagal collapse

Ages: 55 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-09; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of JNJ-54861911 | Pre-dose; 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post-dose on Day 1 of each period
  The Cmax is the maximum observed plasma concentration of JNJ-54861911.
Time to Reach the Maximum Plasma Concentration (Tmax) of JNJ-54861911 | Pre-dose; 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post-dose on Day 1 of each period
  The Tmax is the time to reach the maximum observed plasma concentration of JNJ-54861911.
Area Under the Plasma Concentration-Time Curve From 0 to t Hours (AUC[0-t]) Post Dose of JNJ-54861911 | Pre-dose; 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post-dose on Day 1 of each period
  The AUC (0-t) calculated by trapezoidal summation [time t is the time of the last quantifiable concentration (C[last])].
Area Under the Plasma Concentration-Time Curve From 0 to Infinite Time (AUC[0-infinity]) Post Dose of JNJ-54861911 | Pre-dose; 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post-dose on Day 1 of each period
  The AUC (0-infinity) is the area under the plasma JNJ-54861911concentration-time curve from time 0 to infinite time, calculated as the sum of AUC (0-last) and C(last)/lambda(z), in which AUC(0-last) is area under the plasma JNJ-54861911 concentration-time curve from time zero to time of the last quantifiable concentration, C(last) is the last observed quantifiable concentration and lambda(z) is elimination rate constant.
Elimination Rate Constant (Lambda [z]) of JNJ-54861911 | Pre-dose; 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post-dose on Day 1 of each period
  The Lambda (z) determined by linear regression of the terminal points of the ln-linear plasma concentration-time curve.
Terminal Half-life (t[1/2]) of JNJ-54861911 | Pre-dose; 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post-dose on Day 1 of each period
  The t(1/2) is defined as 0.693/Lambda (z).
Relative Bioavailability (F[rel]) of JNJ-54861911 | Pre-dose; 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post-dose on Day 1 of each period
  Relative bioavailability, calculated as individual Cmax and AUC treatment ratios (for the comparison of food effect).
Rate of Absorption of JNJ-54861911 | Pre-dose; 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post-dose on Day 1 of each period
  Rate of absorption will be measured using the peak concentration of JNJ-54861911 (following administration of solid dosage form and suspension dosage form) under fasted conditions and fed conditions.
Extent of Absorption of JNJ-54861911 | Pre-dose; 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post-dose on Day 1 of each period
  Extent of absorption will be measured under fasted conditions and fed conditions, using the area under plasma concentrations of JNJ-54861911 versus time from time 0 to the last sample point (AUC[0-t]) and from time 0 to infinity (AUC[0-inf]).

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) and Serious AEs | Screening up to follow-up (7 to 14 days after last dose administration)
  An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Merksem, Belgium